CLINICAL TRIAL: NCT00656474
Title: Double-blind, Randomized, Placebo-controlled Phase 2 Pilot Study to Investigate the Safety and Clinical Outcomes of 1.0 % Topically Applied GLYC-101, Compared to Placebo, in Healthy Subjects Undergoing Retro-auricular Carbon Dioxide Laser Skin Resurfacing.
Brief Title: Efficacy Study of GLYC-101 to Evaluate Outcomes After Post-laser Ablation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLYC-101-1a
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Wounds
Keywords: burn wounds; wound healing
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): GLYC-101 Active Retro-auricular Site (1 per participant)
  Interventions: Drug: GLYC-101 gel (1.0 %)
- 2 Comparator (Placebo Comparator): Placebo Retro-auricular Site (1 per participant)
  This arm undergoes laser ablation with subsequent Placebo gel administration
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Placebo gel — Administration of Placebo gel on Day 1, 3 and 5 post ablation.
  Arms: 2 Comparator
Drug: GLYC-101 gel (1.0 %) — Administration on Day 1, 3 and 5 post laser ablation.
  Arms: 1

SUMMARY:
Study is intended to evaluate safety and efficacy parameters in patients treated with GLYC-101 gel or placebo after laser ablation.

DETAILED DESCRIPTION:
The proposed pilot-study will document feasibility, safety and efficacy of topically applied Glucoprime gel (GLYC-101 gel 1.0 %) in promoting wound healing in healthy volunteer subjects undergoing retro-auricular Carbon Dioxide Laser Skin Resurfacing (CO2 LSR). The study will observe the effects of the topical agent over the course of 1 month following the treatment. as a preparation for study GLYC-101-1b (Double-blind, randomized, placebo-controlled Phase 2 Pilot Study to investigate the safety and efficacy of 1.0 % topically applied GLYC 101 compared to placebo, in patients undergoing Carbon Dioxide Laser Skin Resurfacing).

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the study:

* Patients giving informed consent for retro-auricular laser ablation between 25 and 55 years old.
* Retro-auricular area is free of any irritation, scars or dermatologic conditions which might interfere with the study.
* Willing and able to participate in the study and follow all study directions.
* Able to read, understand and sign the consent form.

Exclusion Criteria:

* Pregnant, nursing, or planning a pregnancy during the course of the study, as determined by the interview and a urine pregnancy test.
* Systemic or cutaneous disease that may interfere with the study results.
* Presence of irritation or dermatologic skin conditions in the retro-auricular area.
* Known allergies to materials within the test formulations.
* Systemic or cutaneous therapy with medication that impacts wound healing (steroids, immune modulators, immune suppressants).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph, MD, Principal Investigator — CLINICAL TESTING CENTER of BEVERLY HILLS
Locations (1):
- CLINICAL TESTING CENTER of BEVERLY HILLS, Beverly Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in March 2008 at a single site, Clinical Testing Center of Beverly Hills, Beverly Hills, California, United States, 90210.
Pre-assignment Details: All subjects needed to meet specific inclusion and exclusion criteria as described in the Eligibility section. Eligible subjects were randomly assigned to receive GLYC-101, 1% or placebo.
Groups:
- GLYC-101 and Placebo: Subjects were randomized to receive GLYC-101 Active gel (1%) on one retro-auricular site and Placebo gel on the opposite retro-auricular site.
  GLYC-101 gel (1%) Administration on Day 1, 3 and 5 post laser ablation
Period: Overall Study
Arm/Group | GLYC-101 and Placebo
Started | 12
Completed | 11
Not Completed | 1
Not completed — Other Reason | 1

BASELINE CHARACTERISTICS:
Groups:
- GLYC-101 and Placebo: Subjects were randomized to receive GLYC-101 Active gel (1%) on one retro-auricular site and Placebo gel on the opposite retro-auricular site.
Arm/Group | GLYC-101 and Placebo
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Wound Closure (Epithelialization)
Description: Subjects were evaluated every 2 days from the time of the laser procedures for the first 10 days and then seen every 2 weeks for 4 weeks. Efficacy was assessed based on the time to complete epithelialization in terms of the number of days from Day 1 (day of laser ablation) to the day on which complete epithelialization was observed.
Time Frame: Over the course of 1 month following the initial treatment.
Population: Analysis was Per Protocol.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- GLYC-101 Active Retro-auricular Site (1 Per Participant): GLYC-101 gel (1%) Administration on Day 1, 3 and 5 post laser ablation
- Placebo Retro-auricular Site (1 Per Participant): Placebo gel Administration on Day 1, 3 and 5 post laser ablation
Arm/Group | GLYC-101 Active Retro-auricular Site (1 Per Participant) | Placebo Retro-auricular Site (1 Per Participant)
Number analyzed (Participants) | 12 | 12
days | 15 [15 to 15] | 15 [15 to 15]

2. Secondary Outcome: Percentage of Wound Epithelialized
Description: The percentage of wound epithelialized was assessed at Day 15 post laser ablation.
Time Frame: Day 15 post laser ablation.
Population: Analysis was Per Protocol.
Measure: Number; unit: percent
Arm/Group | GLYC-101 Active Retro-auricular Site (1 Per Participant) | Placebo Retro-auricular Site (1 Per Participant)
Number analyzed (Participants) | 12 | 12
percent | 100 | 100

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the course of 1 month.
Description: AEs were collected at baseline and each study visit.
Arm/Group | GLYC-101 and Placebo
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLYC-101 and Placebo (N=12)
Ear Pruritus (Ear and labyrinth disorders) | 3 (6)
Granuloma (General disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (21)
Erythema (Skin and subcutaneous tissue disorders) | 12 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to 90 days. The sponsor can require changes to the communication to remove any confidential information.